CLINICAL TRIAL: NCT05790070
Title: The Potential Synergistic Effect of Combined Blood Flow Restriction Training and Betaine Supplementation on Skeletal Muscle Mechanotransduction-Associated Cell Signaling
Brief Title: Potential Synergistic Effect of Combined Blood Flow Restriction Training and Betaine Supplementation on Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1676709-6
Record Dates: First submitted 2022-10-20; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Blood Flow Restriction Training; Betaine Supplementation
MeSH Terms: interventions — Betaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 3g/ twice daily (separated by ~12 hours) cellulose placebo for 14 days
  Interventions: Other: Placebo
- Betaine Supplementation (Experimental): 3g/twice daily (separated by ~12 hours) betaine anhydrous for 14 days
  Interventions: Dietary Supplement: Betaine

INTERVENTIONS:
Dietary Supplement: Betaine — 3g/ twice daily (separated by ~12 hours) betaine anhydrous
  Arms: Betaine Supplementation
Other: Placebo — 3g/ twice daily (separated by ~12 hours) cellulose placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether there is a synergistic effect via combining both low-load blood flow restriction (BFR) training and betaine supplementation loading (6g/day for 14 days) on skeletal muscle anabolic signaling pathways that is mediated by enhancements in intracellular water. These effects are proposed to be greater than either BFR training or betaine supplementation alone or compared to control conditions (high-load non-occluded and/or placebo supplementation).

DETAILED DESCRIPTION:
The purpose of the investigation is to determine whether the combination of blood flow restriction (BFR) training and betaine supplementation can synergistically augment phosphorylated targets associated with mechanotransduction and/or muscle protein synthesis relative to either modality alone and compared against control conditions (standard "high-intensity" resistance training and placebo supplementation) in healthy young males. Secondly, the investigators aim to determine if any potential synergistic effects are mediated by enhanced intracellular fluid volumes, as determined by the changes in water content between hydrated and dehydrated muscle samples, as well as through changes in both muscle and serum betaine concentrations. Finally, the investigators aim to assess differences in the aforementioned interventions on specific gene targets, the betaine/γ-aminobutyric acid transporter, myosin heavy chain I, IIa, and IIx lactate dehydrogenase A. Therefore, the specific aims of this study are to determine in healthy, young males: 1) whether combined BFR training and betaine supplementation significantly augment mechanotransductive growth-associated post-translational protein modifications via extra-to-intracellular fluid flux, alongside 2) potentially altered gene expression that otherwise characterizes phenotypical/biochemical changes in skeletal muscle.

The specific aims of the study are to determine whether:

1. The combination of BFR training and betaine supplementation demonstrates significantly greater phosphorylated FAK, ERK1/2, IRS1, and p70S6K, commensurate with greater wet-to-dry hydration changes, relative to any other combinations between BFR training, standard "high-load" training, betaine supplementation, and/or placebo ingestion.
2. The combination of BFR training and betaine supplementation will result in increased MYH2 gene expression, alongside decreases in MYH7 and MYH1 expression. Furthermore, this combination will also result in the highest degree of HIF-1 and Ldha, as well as the lowest BGT-1 gene expression relative to baseline levels.
3. The combination of BFR training and betaine supplementation will result in a higher load-volume accumulated relative to BFR-alone, and will not be statistically different than high-load-placebo training. Therein, the high-load-betaine group will have the greatest load-volume amidst any other combination of conditions.

ELIGIBILITY:
Inclusion Criteria:

* Only participants considered low risk for cardiovascular disease with no contraindications to exercise as outlined by the ACSM
* Have not consumed any nutritional supplements (aside from a multi-vitamin) one month prior to investigation
* Blood pressure <140/90mmHg
* Resting heart rate <90bpm-

Exclusion Criteria:

* sedentary individual as defined by the ACSM guidelines.
* inadequate resistance training experience (<12 months, <3x/week)
* vegetarian, vegan, or have dietary restrictions or supplements that potentially affect betaine metabolism.
* allergy to topical anesthetics.
* known metabolic or cardiovascular disorder including heart disease, arrhythmias, diabetes, thyroid disease, or hypogonadism.
* genetic disorders/polymorphisms that would act as direct contraindications to betaine supplementation (i.e. methyltetrahydrofolate reductase, hyperhomocysteinemia, etc.)
* bleeding disorder, history of pulmonary disease, hypertension, hepatorenal disease, musculoskeletal disorders, neuromuscular/ neurological diseases, autoimmune disease, cancer, peptic ulcers, anemia, or chronic infection (e.g., HIV).
* resting systolic/diastolic blood pressure and heart rate of more than 140/90 mmHg and 90, respectively.
* taking any blood thinning (e.g., warfarin, Jantoven, etc.), heart, pulmonary, thyroid, anti-hyperlipidemic, hypoglycemic, anti-hypertensive, endocrinologic (e.g, thyroid, insulin, etc), emotional/psychotropic (e.g., Prednisone, Ritalin, Adderall), or neuromuscular/neurological medications.
* taking anabolic androgenic steroids within the past year.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
serum/muscle phosphorylated FAK | 3 hours following exercise cessation
  Focal adhesion kinase
insulin receptor substrate 1 | 3 hours following exercise cessation
  signalling adapter protein
gene expression of HIF-1 | 3 hours following exercise cessation
  genes related to skeletal muscle adaptation
serum and muscle betaine concentrations | 3 hours following exercise cessation
  measure related to the supplementation protocol
gene expression BGT-1 | 3 hours following exercise cessation
  genes related to skeletal muscle adaptation
gene expression MHC | 3 hours following exercise cessation
  genes related to skeletal muscle adaptation

SECONDARY OUTCOMES:
pre-to-post exercise set tissue hydration | both pre and immediately post exercise session
  hydration status of the participant via multi-frequency bioelectrical impedance
capillary blood lactate concentrations | both pre and immediately post exercise session
  blood lactate levels of the participant
set-to-failure repetition number | immediately post exercise session
  as related to the exercise protocol
exercise condition total load-volume. | immediately post exercise session
  as related to the exercise protocol and calculated at termination of the exercise session

CONTACTS AND LOCATIONS:
Overall Officials: LesLee Funderburk, PhD, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No